CLINICAL TRIAL: NCT05231616
Title: Magnetic Resonance Imaging Based Deep Learning Model for Diagnosis and Contour of Cervical Lymph Node for Nasopharyngeal Carcinoma: a Multicenter Study
Brief Title: Deep Learning Model for Diagnosis and Contour of Cervical Lymph Node for Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Professor, Sun Yat-sen University
Other Study IDs: B2020-334
Record Dates: First submitted 2022-02-08; First posted 2022-02-09 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Deep Learning Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnosis of cervical lymph node in nasopharyngeal carcinoma is difficult. Magnetic resonance imaging based deep learning model may be a noninvasive and rapid diagnostic method for cervical lymph node. Thus, the investigators aimed to develop and externally validate a deep learning model to assist in the diagnosis and localization of metastatic lymph nodes in nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of nasopharyngeal carcinoma; Cervival lymph nodes confirmed by pathology

Exclusion Criteria:

* a history of cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nasopharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | 2022-12-31

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China